CLINICAL TRIAL: NCT01243463
Title: Effects of Bariatric Surgery on Obstructive Sleep Apnea
Brief Title: Bariatric Surgery and Obstructive Sleep Apnea
Acronym: BAROSA
Status: Completed | Type: Observational
Sponsor: Summa Health System (Other)
Responsible Party: Rachael Pohle-Krauza, Summa Health System
Other Study IDs: RP09125
Record Dates: First submitted 2010-11-16; First posted 2010-11-18 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Obstructive Sleep Apnea; Bariatric Surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
More often than not, obesity occurs in tandem with Obstructive Sleep Apnea (OSA), and each disease effectively perpetuates severity of the other. Surgical weight loss (i.e. bariatric surgery), and nocturnal, positive airway pressure therapy (PAP) are used to treat the two conditions separately, and these treatment modalities both present a unique set of challenges in terms of patient-adherence. Furthermore, the combined effects of these therapies on body weight and OSA severity are unclear, and require longitudinal investigation. The purpose of the research proposed herein is twofold: A) To prospectively demonstrate the specific physiologic/psychological improvements in OSA risk factors and disease severity that occur in a subset of bariatric surgery patients with OSA, who are being effectively treated with PAP and furthermore; B) To elucidate differences in postoperative outcomes (weight-loss, dyslipidemia, OSA severity, comorbidity resolution) between patients who are compliant or non-compliant with prescribed PAP therapy. The investigators anticipate that results will be used to develop and streamline approaches to improve pulmonary/sleep-related outcomes in bariatric surgery patients. Furthermore, this line of research has many implications for strategies to strengthen the coordination of care between bariatric surgery, pulmonology, and other clinical sub-specialties that are integral to the postoperative health of these patients.

ELIGIBILITY:
Inclusion Criteria:

* obese (Body Mass Index > 35)
* pending laparoscopic roux-en-Y gastric bypass at Summa Bariatric Care Center
* women
* ages 20 - 85
* diagnosed OSA and prescribed nocturnal, autotitrating positive airway pressure therapy

Exclusion Criteria:

* are excluded if failure to meet any of the above

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese women, 20 - 85 years of age
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-02

CONTACTS AND LOCATIONS:
Locations (1):
- Summa Health System Akron City Hospital, Akron, Ohio, United States